CLINICAL TRIAL: NCT04168372
Title: Fructose: Substrate, Stimulus, or Both?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Touro University, California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: M-3018
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Insulin Resistance; Insulin Sensitivity; Pre Diabetes
Keywords: Fructose; Glucose; Lipogenesis
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High fructose meal, with fructose label (Experimental): 2-13C fructose incorporated into a meal with high fructose content
  Interventions: Other: High fructose, fructose labeled meal
- High fructose meal, with pyruvate label (Experimental): 2-13C pyruvate incorporated into a meal with high fructose content
  Interventions: Other: High fructose, pyruvate labeled meal
- Low fructose meal, with fructose label (Experimental): 2-13C fructose incorporated into a meal with low fructose content
  Interventions: Other: Low fructose, fructose labeled meal
- Low fructose meal, with pyruvate label (Experimental): 2-13C pyruvate incorporated into a meal with low fructose content
  Interventions: Other: Low fructose, pyruvate labeled meal

INTERVENTIONS:
Other: High fructose, fructose labeled meal — Liquid meal containing high fructose (16% of energy), labeled with 2-13C fructose
  Arms: High fructose meal, with fructose label
Other: High fructose, pyruvate labeled meal — Liquid meal containing high fructose (16% of energy), labeled with 2-13C pyruvate
  Arms: High fructose meal, with pyruvate label
Other: Low fructose, fructose labeled meal — Liquid meals containing low fructose (6% of energy), labeled with 2-13C fructose
  Arms: Low fructose meal, with fructose label
Other: Low fructose, pyruvate labeled meal — Liquid meal containing low fructose (6% of energy), labeled with 2-13C pyruvate
  Arms: Low fructose meal, with pyruvate label

SUMMARY:
This objective of this study is to use sensitive methodology under controlled conditions to investigate the mechanisms by which fructose consumption contributes to excess fatty acid synthesis and elevations in blood glucose levels following consumption of meals containing fructose.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index 22 to 35 kg/m2
* Prediabetic (HbA1c 5.7% to 6.5%) or hyperinsulinemic (fasting insulin ≥12 µIU/mL) but non-diabetic (fasting glucose <126mg/dL and HbA1c < 6.5%) ; or normal control (fasting insulin <10 µIU/mL, fasting glucose <100 mg/dL, and HbA1c < 5.7%)

Exclusion Criteria:

* Pregnancy or lactation within the past six months
* Type 1 or 2 diabetes mellitus
* History of liver disease or aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 2x the upper limit of normal (ULN);
* Fasting triglyceride or total cholesterol levels above 95th percentile for age and sex;
* Hemoglobin or hematocrit below the lower limit of normal for sex;
* Report of hepatitis or HIV infection;
* History of cancer, use of any anti-diabetic medications or hypolipidemic agents in the past six months;
* History of surgical procedure for obesity;
* Self-reported change in body weight >5% in the past six months;
* History of other conditions known to affect insulin sensitivity and lipid metabolism;
* Known intolerance to acetaminophen or components of the liquid test meals.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Hepatic fractional de novo lipogenesis in triglyceride rich lipoprotein (TRL) | 6 hours
  Measured by the detection of 13C carbons in TRL-palmitate from administered 13C labeled pyruvate or 13C labeled fructose.
Rate of appearance of UDP-glucose | 6 hours
  An estimate of hepatic glycogen flux measured by administration of D1 galactose and acetaminophen
Rate of appearance of blood glucose from gluconeogenesis | 6 hours
  Measured by the dilution method of labeled glucose

SECONDARY OUTCOMES:
Serum triglyceride concentration | 6 hours
  Fasting and postprandial serum triglyceride levels
Serum glucose concentration | 6 hours
  Fasting and postprandial serum triglyceride levels
Serum lactate concentration | 6 hours
  Fasting and postprandial serum lactate levels
Serum insulin concentration | 6 hours
  Fasting and postprandial insulin levels
Serum free fatty acid concentration | 6 hours
  Fasting and postprandial fatty acid levels
Enteral (chylomicron) fractional de novo lipogenesis (DNL) | 6 hours
  Measured by the detection of 13C carbons in chylomicron-palmitate from administered 13C labeled pyruvate or 13C labeled fructose.
Hepatic (VLDL) fractional de novo lipogenesis (DNL) | 6 hours
  Measured by the detection of 13C carbons in VLDL-palmitate from administered 13C labeled pyruvate or 13C labeled fructose.
Extrasplanchnic fructose | 6 hours
  Calculated using total plasma fructose, plasma 2-13C fructose enrichment, and endogenous fructose production
Whole body fructose oxidation | 6 hours
  Measured by 13C atom % excess in exhaled breath, and VCO2 by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Schwarz, PhD, Principal Investigator — Touro University, California
Locations (1):
- Touro University California, Vallejo, California, United States

IPD SHARING:
Plan to Share IPD: No